CLINICAL TRIAL: NCT05055635
Title: ReRad III. Pencil Beam Proton Therapy for Recurrences in Anal Cancer Patients Previously Treated With Radiotherapy
Brief Title: Pencil Beam Proton Therapy for Recurrences in Anal Cancer Patients Previously Treated With Radiotherapy (DACG 5)
Acronym: ReRad III
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCPT070721
Record Dates: First submitted 2021-07-08; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-07

CONDITIONS: Anal Cancer; Recurrent Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Doseescalated pencil beam proton therapy (Experimental): Neo-adjuvant or definitive pencil beam proton therapy: 55 Gy(RBE)/44fx - 65 Gy(RBE)/52 fx (1.25 Gy per fraction), two fractions a day.
  Interventions: Radiation: Pencil beam proton therapy

INTERVENTIONS:
Radiation: Pencil beam proton therapy — Neo-adjuvant or definitive pencil beam proton therapy: 55 Gy(RBE)/44fx - 65 Gy(RBE)/52 fx (1.25 Gy per fraction), two fractions a day

SUMMARY:
This protocol aims to determine toxicity and efficacy of re-irradiation for patients with recurrences from anal cancers with dose-escalated pencil beam proton therapy either pre-operative for marginally resectable recurrences or as a definitive treatment strategy (un-resectable, operation declined etc.). The over-all aim is to improve local tumor control with acceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent anal cancer
* Bioptically verified (squamous cell carcinoma)
* Available dose plan from primary radiotherapy
* Previous RT (>30Gy EQD2)
* Evaluated in MDT-conferences (Herlev, Aarhus)
* Age>18 years
* PS 0-2
* Adequate organ function
* Written informed consent

Exclusion Criteria:

* Distant metastases deemed without curative intended treatment options (PET-CT)
* Unable to undergo MRI, PET-CT
* Inability to attend full course radiotherapy and follow up in the outpatient clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2027-07-06 (Estimated); Study Completion 2030-07-06 (Estimated)

PRIMARY OUTCOMES:
Local control | 12 months
  MRI

SECONDARY OUTCOMES:
Local re-recurrence | 6 and 24 months
Progression free survival | 3-5 year FU
Overall survival | 3-5 year FU
Pathological evaluation of R0, R1 or R2 resection | 6 months
Toxicity | up to 6 weeks, 1 year, 3 year
  evaluated by NCI-CTCAE v. 5.0
Quality of life assessment | up to 6 weeks, 1 year, 3 year
  EORTC QLQ-c30
Quality of life assessment | up to 6 weeks, 1 year, 3 year
  QLQ-CR29
Quality of life assessment | up to 6 weeks, 1 year, 3 year
  QLQ-ANL27
Quality of life assessment | up to 6 weeks, 1 year, 3 year
  LARS score
Translational research | baseline, end of therapy, 1 year
  cfDNA
Summed radiotherapy dose volume to organs at risk and correlation to toxicities | up to 6 weeks, 1 year, 3 year
To investigate 30-day surgical overall morbidity | 30-day
  Clavien-Dindo
To investigate 6-month surgical site morbidity | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Centre for Particle Therapy, Aarhus N, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No